CLINICAL TRIAL: NCT01937806
Title: A Phase Ⅲ, Multi-center, Randomized, Double-blinded, Parallel Study to Assess the Antiviral Activity and Safety of Besifovir 150 mg Compared to Tenofovir 300 mg in Chronic Hepatitis B Patients for 48 Weeks
Brief Title: Phase 3 and Extensional Study of Besifovir
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID_BVCL011
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — ((1-((2-amino-9H-purin-9-yl)methyl)cyclopropyl)oxy)methylphosphonic acid dipivoxyl; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- besifovir 150mg (Experimental): Besifovir 150 mg q.d. + Placebo of Tenofovir Disoproxil Fumarate 300 mg q.d. + L-carnitine (L-Carn Tab. 330 mg) 660 mg q.d.
  Interventions: Drug: besifovir 150mg
- Tenofovir 300mg (Active Comparator): Placebo of Besifovir 150 mg q.d. + Tenofovir Disoproxil Fumarate 300 mg q.d. + Placebo of L-carnitine (L-Carn Tab. 330 mg) 660 mg q.d.
  Interventions: Drug: tenofovir 300mg

INTERVENTIONS:
Drug: besifovir 150mg — Besifovir 150 mg q.d. + Placebo of Tenofovir Disoproxil Fumarate 300 mg q.d. + L-carnitine (L-Carn Tab. 330 mg) 660 mg q.d.
  Arms: besifovir 150mg
Drug: tenofovir 300mg — Placebo of Besifovir 150 mg q.d. + Tenofovir Disoproxil Fumarate 300 mg q.d. + Placebo of L-carnitine (L-Carn Tab. 330 mg) 660 mg q.d.
  Arms: Tenofovir 300mg

SUMMARY:
To prove that a study drug is noninferior to a control drug with a proportion of subjects who showed HBV DNA undetected (less than 400 copies/mL (69 IU/mL)) at the 48th week after 48-week administration of Besifovir 150 mg, or Tenofovir 300 mg as a control drug to chronic hepatitis B patients

DETAILED DESCRIPTION:
* Screening Period Subject registration is conducted with confirming selection and exclusion criteria after a written consent form is obtained within 28 days before clinical trial drug administration.
* Wash-out Period Subjects who had been treated with antiviral agents within 12 weeks should complete a 4-week wash-out period from the stage of stopping antiviral agent treatment before a baseline visit and subjects who have no experience of antiviral agent treatment start a baseline visit without a wash-out period.
* Baseline Subjects who visit on the date of starting clinical trial drug administration are randomized to a test group or a control group at a ratio of 1:1. Double blindness is applied for both groups.
* Treatment period Subjects are orally administered with a clinical trial drug q.ds.i.d. for 48 weeks and visit at the 0, 4th, 12th, 24th, 36th, and 48th week for an HBV DNA test, laboratory tests, a physical test, vital signs, and adverse events.
* Follow-up period Subjects are provided with appropriate treatment after completing the 48-week trial or dropping out. Subjects visit once at the 60th week for follow-up of adverse events, such as acute deterioration of hepatitis B, and HBV DNA test results. If any treatment is not conducted after 48-week administration, subjects visit at intervals of four weeks until a follow-up visit (60th week) and the same tests with the 24th week visit (Visit 5) are conducted. However, subjects who participate in a 48-week separate extended trial conducted after 48-week administration in this clinical trial do not have a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients over the age of 20 years old
2. Patients who show positive HBsAg or has a history of chronic hepatitis B for the last six months or more before screening
3. Patients who have not received interferon (including Pegylation formulation) to treat chronic hepatitis and antiviral agents for more than 12 weeks.
4. Patients who showed positive HBsAg during screening
5. Patients who showed HBV DNA measured by COBAS TaqManTM HBV Test more than 1x105 copies/mL (17,241 IU/mL) in case of positive HBeAg during screening, or who showed HBV DNA measured by COBAS TaqManTM HBV Test more than 1x104 copies/mL (1,724 IU/mL) in case of negative HBeAg
6. Patients who showed ALT more than 1.2 times, or less than 10 times of the upper limit in the normal range during screening
7. Patients who were explained about the purpose, methods and effects of the clinical trial and then, signed a written consent form.
8. Male and female patients of childbearing age who can use double contraception acknowledged* during a trial period * Double contraception acknowledged means combination of barrier contraception (condom, diaphragm, etc.) and other contraception (sterilization operation, intrauterine contraceptive device, oral contraceptive drug, other hormone delivery system, contraceptive cream, jelly or foam, etc.).

Exclusion Criteria:

1. Patients who have hepatitis C (HCV), hepatitis D (HDV), or human immunodeficiency virus (HIV)
2. Patients with a uncompensated liver disease who have at least one of the following values or signs during screening

   * Total bilirubin > 2 x ULN
   * Prothrombin time delayed more than three seconds compared to the normal value
   * Serum Albumin < 30 g/L (3 g/dL)
   * A medical history of ascites, jaundice, hemorrhage by varix, hepatic encephalopathy, or other signs of liver function loss
3. At least one of the following laboratory values during screening

   * Hemoglobin < 9.0 g/dL
   * Absolute neutrophil count (ANC) < 1.5 x 109 /L (1500 /mm3)
   * Platelet count < 100 x 109 /L (100 x 103 /mm3)
   * Serum creatinine > 1.5 mg/dL
   * Serum amylase > 2 x ULN and Lipase > 2 x ULN
4. Patients who showed GFR less than 50 mL/min by calculating MDRD (Modification of Diet in Renal Disease: 1.86 x PCr -1.154 x AGE -0.203 (x 0.742 for women)) during screening
5. Patients who showed alpha-fetoprotein(AFP) more than 50 ng/mL during screening and are estimated to have hepatocellular carcinoma (HCC) through liver/abdomen CT scans
6. Patients who had received the following drugs for the last two months before screening (however, short-term use (less than consecutive 14 days) of these drugs and low-dose aspirin (100 mg, maximally, 300 mg/day) are allowed.)

   * Nephrotoxic drugs (e.g. Aminoglycosides, Amphotericin B, NSAIDs)
   * Hepatotoxic drugs (e.g. Erythromycin, Ketoconazole, Rifampin, Fluconazole, Dapsone)
   * Anticoagulant (e.g. Warfarin)
7. Patients who are suspected by an investigator to have the level of immunity decreased among patients who had been administered with immunosuppressants within six months before screening
8. Patients who had been administered with long-term general corticosteroids (more than consecutive 14 days) at a high dose (more than prednisolone 20 mg daily*) within three months before screening (In case of local corticosteroids, an investigator decides it.)

   * It is equal to cortisone 125 mg, hydrocortisone 100 mg, prednisone 20 mg, methylprednisolone 16 mg, triamcinolone 16 mg, dexamethasone 3 mg, betamethasone 2.4 mg.
9. Patients who were diagnosed as a malignant tumor within five years before screening or have a relapse of a malignant tumor (In case of a benign tumor, if an investigator decides that it does not affect the progress of the clinical trial during a trial period, the patients can be registered.)
10. Patients who are scheduled to participate in other clinical trial after registered in this clinical trial, or had been participated in other clinical trial within three months before registered in this clinical trial
11. Pregnant women, lactating women, or patients who planned pregnancy during a trial period
12. Patients who have hypersensitivity to the clinical trial drug in this clinical trial
13. Patients who have a past medical history of clinical alcohol or drug abuse within a year before screening or now are abusers
14. Patients who have a severe disease, such as liver diseases, heart failure, renal failure, and pancreatitis, decided by an investigator to have an effect on this clinical trial
15. Patients who have other hepatic diseases (hematochromatosis, Wilson's disease, alcoholic liver diseases, nonalcoholic steatohepatitis, α1-antitrypsin deficiency) except hepatitis B
16. Patients who received an organ transplant
17. Persons who are possible to decline daily function due to a mental disease or patients who are not able to understand the purpose and methods of this clinical trial
18. Patients who are decided by an investigator as unsuitable for conducting this clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
The rate of subjects who showed HBV DNA undetected (less than 400 copies/mL (69 IU/mL)) at the 48th week | at the 48th week
  The rate of subjects who showed HBV DNA undetected (less than 400 copies/mL (69 IU/mL)) at the 48th week

SECONDARY OUTCOMES:
The rate of subjects who showed HBV DNA less than 116 copies/mL (20 IU/mL, LOQ of COBAS TaqManTM) at the 48th week | at the 48th week
  The rate of subjects who showed HBV DNA less than 116 copies/mL (20 IU/mL, LOQ of COBAS TaqManTM) at the 48th week
Average amount of change in an HBV DNA common logarithm value at the 48th week to a base value | at the 48th week
  Average amount of change in an HBV DNA common logarithm value at the 48th week to a base value
The rate of subjects who showed ALT normalized at the 48th week | at the 48th week
  The rate of subjects who showed ALT normalized at the 48th week
The rate of subjects who showed HBV DNA undetected (less than 400 copies/mL (69 IU/mL)) and ALT normalized at the 48th week | at the 48th week
  The rate of subjects who showed HBV DNA undetected (less than 400 copies/mL (69 IU/mL)) and ALT normalized at the 48th week
The rate of subjects who showed HBsAg serum loss and/or seroconversion (HBsAg loss and Anti-HBs formation) at the 48th week | at the 48th week
  The rate of subjects who showed HBsAg serum loss and/or seroconversion (HBsAg loss and Anti-HBs formation) at the 48th week
The rate of subjects who showed HBeAg serum loss and/or seroconversion (HBeAg loss and Anti-HBe formation) at the 48th week among subjects with positive HBeAg | at the 48th week
  The rate of subjects who showed HBeAg serum loss and/or seroconversion (HBeAg loss and Anti-HBe formation) at the 48th week among subjects with positive HBeAg
The rate of subjects who showed HBV DNA undetected (less than 400 copies/mL (69 IU/mL)) and HBeAg loss at the 48th week among subjects with positive HBeAg | at the 48th week
  The rate of subjects who showed HBV DNA undetected (less than 400 copies/mL (69 IU/mL)) and HBeAg loss at the 48th week among subjects with positive HBeAg
The rate of subjects who showed HBV DNA undetected (less than 400 copies/mL (69 IU/mL)) and HBeAg seroconversion at the 48th week among subjects with positive HBeAg | at the 48th week
  The rate of subjects who showed HBV DNA undetected (less than 400 copies/mL (69 IU/mL)) and HBeAg seroconversion at the 48th week among subjects with positive HBeAg
Changes in antiviral drug resistant mutation according to HBV DNA sequencing results at the 48th week | at the 48th week
  Changes in antiviral drug resistant mutation according to HBV DNA sequencing results at the 48th week
The rate of subjects who showed virologic breakthrough according to serum HBV DNA at the 48th week | at the 48th week
  The rate of subjects who showed virologic breakthrough according to serum HBV DNA at the 48th week

CONTACTS AND LOCATIONS:
Overall Officials: Kwan Sik Lee, M.d., Ph.D, Principal Investigator — Kangnam Severance Hospital, Yonsei University, Seoul, Korea; Young Oh Kweon, M.D., Ph.D, Principal Investigator — Kyungpook National University Hospital, Seoul, Korea; Hyung Joon Yim, M.D., Ph.D., Principal Investigator — Korea University Medical Center, Ansan, Kyunggi-do, Korea; Soon Ho Um, M.D., Ph.D., Principal Investigator — Korea University Medical Center, Seoul, Korea; Won Kim, M.D., Ph.D., Principal Investigator — Seoul National University Boramae medical Center, Seoul, Korea; Sung Jae Park, M.D., Ph.D., Principal Investigator — Inje University Busan Paik Hospital, Pusan, Korea; Yoon Jun Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital, Seoul, Korea; Yoon Jun Kim, M.D., Ph.D., Principal Investigator — The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Korea; Young-Suk Lim, M.D., Ph.D., Principal Investigator — Asan Medical Center, Seoul, Korea; JinMo Yang, M.D., Ph.D., Principal Investigator — The Catholic University of Korea, Seoul St. Vincent's Hospital, Seoul, Korea; Jang, Jae Young, M.D., Ph.D., Principal Investigator — Soonchunhyang University Hospital, Seoul, Korea; Jae-Youn Cheong, M.D., Ph.D., Principal Investigator — Ajou University Medical Center, Suwon, Kyunggi-do, Korea; Neung Hwa Park, M.D., Ph.D., Principal Investigator — Ulsan University Hospital, Ulsan, Korea; Moon Young Kim, M.D., Ph.D., Principal Investigator — Wonju Sevrerance Christian Hospital, Wonju, Kangwon-do, Korea; Jin-Woo Lee, M.D., Ph.D., Principal Investigator — Inha University Hospital, Incheon, Inchen, Korea; Dong Joon Kim, M.D., Ph.D., Principal Investigator — Hallym University Medical Center, ChunCheon, Kangwon-do, Korea; Byung Seok Lee, M.D., Ph.D., Principal Investigator — Chungnam National University Hospital; Joo Hyun Sohn, M.D., Ph.D., Principal Investigator — Hanyang University Guri Hospital, Guri, Kyunggi-do, Korea; Kwang-Hyub Han, M.D., Ph.D., Principal Investigator — Severance Hospital of Yonsei University, Seoul, Korea; Hong Soo Kim, M.D., Ph.D., Principal Investigator — Soonchunhyang University Hospital, Choenan, Chungchoengnam-do, Korea
Locations (20):
- South Korea (20):
  - Soonchunhyang University Hospital, Cheonan, Chungchoengnam-do
  - Hallym University Medical Center, Chuncheon, Gangwon-do
  - Wonju Sevrerance Christian Hospital, Wŏnju, Gangwon-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Ajou University Medical Center, Suwon, Gyeonggi-do
  - Korea University Medical Center, Ansan, Kyounggi-do
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Inha University Hospital, Incheon
  - Inje University Busan Paik Hospital, Pusan
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Medical Center, Seoul
  - Seoul National University Boramae medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital of Yonsei University, Seoul
  - Soonchunhyang University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Vincent's Hospital, Seoul
  - Ulsan University Hospital,, Ulsan

REFERENCES:
- [Derived] Yim HJ, Kang SH, Jung YK, Ahn SH, Kim W, Yang JM, Jang JY, Kweon YO, Cho YK, Kim YJ, Hong GY, Kim DJ, Sohn JH, Lee JW, Park SJ, Yim SY, Park JK, Um SH. Reduced Risk of Hepatocellular Carcinoma in Patients with Chronic Hepatitis B Receiving Long-Term Besifovir Therapy. Cancers (Basel). 2024 Feb 22;16(5):887. doi: 10.3390/cancers16050887. PMID 38473248
- [Derived] Song DS, Kim W, Ahn SH, Yim HJ, Jang JY, Kweon YO, Cho YK, Kim YJ, Hong GY, Kim DJ, Jung YK, Sohn JH, Lee JW, Park SJ, Lee BS, Kim JH, Kim HS, Yoon SK, Kim MY, Lee KS, Lim YS, Lee WS, Yang JM, Kim KH, Han KH, Um SH. Continuing besifovir dipivoxil maleate versus switching from tenofovir disoproxil fumarate for treatment of chronic hepatitis B: Results of 192-week phase 3 trial. Clin Mol Hepatol. 2021 Apr;27(2):346-359. doi: 10.3350/cmh.2020.0307. Epub 2021 Jan 25. PMID 33493393
- [Derived] Yim HJ, Kim W, Ahn SH, Yang JM, Jang JY, Kweon YO, Cho YK, Kim YJ, Hong GY, Kim DJ, Jung YK, Um SH, Sohn JH, Lee JW, Park SJ, Lee BS, Kim JH, Kim HS, Yoon SK, Kim MY, Lee KS, Lim YS, Lee WS, Han KH. Besifovir Dipivoxil Maleate 144-Week Treatment of Chronic Hepatitis B: An Open-Label Extensional Study of a Phase 3 Trial. Am J Gastroenterol. 2020 Aug;115(8):1217-1225. doi: 10.14309/ajg.0000000000000605. PMID 32355123
- [Derived] Ahn SH, Kim W, Jung YK, Yang JM, Jang JY, Kweon YO, Cho YK, Kim YJ, Hong GY, Kim DJ, Um SH, Sohn JH, Lee JW, Park SJ, Lee BS, Kim JH, Kim HS, Yoon SK, Kim MY, Yim HJ, Lee KS, Lim YS, Lee WS, Park NH, Jin SY, Kim KH, Choi W, Han KH. Efficacy and Safety of Besifovir Dipivoxil Maleate Compared With Tenofovir Disoproxil Fumarate in Treatment of Chronic Hepatitis B Virus Infection. Clin Gastroenterol Hepatol. 2019 Aug;17(9):1850-1859.e4. doi: 10.1016/j.cgh.2018.11.001. Epub 2018 Nov 15. PMID 30448598